CLINICAL TRIAL: NCT02930811
Title: Efficacy of Sildenafil on the Morbi-mortality of Peripheral Arterial Diseased Patients With Intermittent Claudication. A National, Multicentre, Prospective, Randomised, Double-Blind, Placebo-Controlled Trial.
Brief Title: Efficacy of Sildenafil on the Morbi-mortality of Peripheral Arterial Diseased Patients With Intermittent Claudication
Acronym: VALSTAR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Investigator-Coordinator has moved to Rennes University Hospital. It will be done under the sponsor of Rennes University Hospital : NCT03686306
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC-N-2015
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil (Experimental): Single Sildenafil oral morning intake (100mg/day) per day for a total duration of 6 months (Sildenafil 100 mg oral morning dose)
  Interventions: Drug: Sildenafil 100 mg oral morning dose
- Placebo (Placebo Comparator): Single Placebo oral morning intake per day for a total duration of 6 months (Placebo oral morning dose)
  Interventions: Drug: Placebo oral morning dose

INTERVENTIONS:
Drug: Sildenafil 100 mg oral morning dose — Measurement of maximal walking distance on a constant load treadmill test, SF-36 questionnaire, and Edimburg questionnaire at inclusion, 1 month, 3 month and 6 month.
  Events occurence questionnaires, Tolerance and adverse events questionnaire, Welch questionnaire and walk recommendation at inclusion, 7 days, 14 days, 1-2-3-4-5-6 and 9 months
  Other Names: Experimental: Sildenafil
  Arms: Sildenafil
Drug: Placebo oral morning dose — Measurement of maximal walking distance on a constant load treadmill test, SF-36 questionnaire, and Edimburg questionnaire at inclusion, 1 month, 3 month and 6 month.
  Events occurence questionnaires, Tolerance and adverse events questionnaire, Welch questionnaire and walk recommendation at inclusion, 7 days, 14 days, 1-2-3-4-5-6 and 9 months
  Other Names: Placebo Comparator: Placebo
  Arms: Placebo

SUMMARY:
Peripheral Arterial Disease (PAD) is a highly debilitating disease that affects 202 million people around the world and about 7 million people in France. Morbi-mortality from cardiovascular events is increased in this population. Intermittent claudication is the most common clinical feature of PAD.

Primary therapeutic approach is medical treatment and advice to walk. Sildenafil, a PDEi type 5, is well tolerated, largely used in impotence and has interesting clinical delay and duration of action in the concept of a potential use in claudication.

For patients agreeing and signing informed consent, randomisation of treatment (placebo/sildenafil) will be done. Treatment will be proposed in addition to usual treatment. The experimental drug will be delivered for a 1 month treatment. First follow up visit at month one will focus on tolerance, compliance and eventual side effects. If no major side effect is found the study drug will then be delivered for an additional 2 months. Patients will be evaluated at month 3 (second follow-up visit) for persistent or non-persistent indication for revascularisation and addressed for revascularization if needed. In parallel focus on tolerance, compliance and eventual side effects will be done. If no major side effect is found, the study drug will be delivered for an additional 3 months treatment. Third and fourth follow-up visit are scheduled at month 6 (end of treatment) and month 9 (3 months after the end of experimental drugs).

ELIGIBILITY:
Inclusion Criteria:

* Grade I cat 2 or 3 claudication despite optimal medical treatment
* Reporting a vascular claudication history for at least 3 months
* Able to achieve a walking treadmill test, Walking time on treadmill (3.2km/h, 10% slope) less than 5 minutes
* Having no cons Sildenafil indication
* Must be on optimal medical therapy (ACE Inhibitors / AT2 Antagonist + Antiplatelet + Lipid Lowering drugs) for at least 1 month

Exclusion Criteria:

* Critical ischemia
* Previous history of myocardial infarction or angina not stabilized
* Amblyopia
* Treated with nitrates (nitroglycerin ...) or drugs interfering with the action of the Sildenafil
* Pregnant woman and woman in labor
* Major Person subject to reinforced protection, deprived of their liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social establishment for purposes other than research
* Being in an exclusion period for another biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of Event free survival rate | 6 months after the treatment begining
  Event free survival is defined as the time between inclusion date and the date of event occurrence. If no event is observed at the follow-up period, event free survival is defined as the delay of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Loukman OMARJEE, MD, Study Director — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omarjee L, Camarzana A, Henni S, Abraham P. Nonrevascularizable buttock claudication improved with Sildenafil: A case report. Medicine (Baltimore). 2017 Feb;96(8):e6186. doi: 10.1097/MD.0000000000006186. PMID 28225505